CLINICAL TRIAL: NCT05462483
Title: Heat Application to the Quadriceps Musculature and Its Effect on Pain Following a Total Knee Arthroplasty
Brief Title: Heat Application to Quadriceps Effect on Pain After a Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Idaho Clinic (Other)
Responsible Party: Principal Investigator, Cole Adams, Principal Investigator, The Idaho Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IdahoClinic
Record Dates: First submitted 2022-05-27; First posted 2022-07-18 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Arthritis Knee

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rice sock and instructions to heat quadriceps (Experimental): Receives heating device and instructions to heat the quadriceps musculature.
  Interventions: Other: Rice Sock and Instructions to heat the quadriceps.
- No heating device or instructions to heat quadriceps (No Intervention): WIll not receive heating device or instructions to heat quadriceps musculature.

INTERVENTIONS:
Other: Rice Sock and Instructions to heat the quadriceps. — A rice sock will be provided to the experimental group to heat the quadriceps 3x per day for six weeks. The participants will be encouraged to heat before and after rehabilitation exercises as well.
  Arms: Rice sock and instructions to heat quadriceps

SUMMARY:
The goal of this study is to explore an under-researched aspect of recovery. Typically, post-operative care after a knee arthroplasty consists of compression (stockings), medications, rest, ice, elevation, physical therapy, and wound care. All of these treatments perform their role well, however, medications such opiates run the risk of addiction. An additional method of pain management such as heat application to the surrounding musculature warrants exploration.

The goal of this study is to reduce the amount of pain, and improve the quality of life in post-operative patients. Pain, stiffness, symptoms, quality of life and function of the knee will be evaluated utilizing patient-reported measures and range of motion. Patients will be assessed using the Knee Injury and Osteoarthritis Outcome survey (KOOS Jr), Visual Analogue Scale (VAS) and PROMIS. Patients will be given these surveys during their two and six week check-in with the surgeon. In addition to these patient-reported measures, the investigators will also be tracking range of motion (ROM) and opioid usage. The data will then be collected via the patient's electronic health record, or by the researcher directly. The treatment group will be given a written order to apply heat to the quadriceps at least three times per day for 10-15 minutes each. This can be done in four hour increments or when patients symptoms begin to worsen. The patient will receive a rice sock for heat application. The control group will not be withheld from heat application, but will not be instructed to do so. The control group will instead follow the current standard of care as advised by the physician.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a total knee arthroplasty ages 18 and older at Saint Alphonsus Hospital and at The Idaho Clinic between the months of June-February, or until the estimated sample size (150) is reached. Must be able to withstand heat to thigh. Must consent to research.

Exclusion Criteria:

* Anyone unable to give informed consent, pregnant individuals, children, or anyone whom the intervention may be harmful to.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Change of Pain experienced at 2 and 6 week check-ins | Baseline, 2, and 6 week evaluations
  Measured via KOOS Jr survey
Change of Pain experienced at 2 and 6 week check-ins | Baseline, 2, and 6 week evaluations
  Measured via VAS survey
Change of Pain experienced at 2 and 6 week check-ins | Baseline, 2, and 6 week evaluations
  Measured via PROMIS survey
Change in stiffness experienced at 2 and 6 week check-ins | Baseline, 2 and 6 week evaluations
  Measured via PROMIS survey
Change in stiffness experienced at 2 and 6 week check-ins | Baseline, 2 and 6 week evaluations
  Measured via KOOS Jr survey
Change in quality of life at 2 and 6 week check-ins | Baseline, 2 and 6 weeks
  Measured via PROMIS survey
Change in Physical Health | Baseline, 2 and 6 weeks
  Measured via PROMIS survey
Change in Mental Health | Baseline, 2 and 6 weeks
  Measured via PROMIS survey
Change in knee function at 2 and 6 week check-ins | Baseline, 2 and 6 weeks
  Measured via Range of motion
Change in knee function at 2 and 6 week check-ins | Baseline, 2 and 6 weeks
  Measured via PROMIS surveys
Change in knee function at 2 and 6 week check-ins | Baseline, 2 and 6 weeks
  Measured via KOOS Jr

SECONDARY OUTCOMES:
Opiate Refills | Up to 6 weeks post-operation
  Opiate usage/refills will be evaluated
Change in Range of Motion at 2 and 6 week check-ins | Baseline, 2 and 6 week check-ins
  ROM will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Cole Adams, Principal Investigator — Idaho College of Osteopathic Medicine
Locations (1):
- The Idaho Clinic, Boise, Idaho, United States

DOCUMENTS (1):
  • Informed Consent Form (2022-07-13): https://cdn.clinicaltrials.gov/large-docs/83/NCT05462483/ICF_000.pdf